CLINICAL TRIAL: NCT01659723
Title: Radiation Induced Cystitis Treated With Hyperbaric Oxygen - A Randomized Controlled Trial
Acronym: RICH-ART
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Sahlgrenska University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RICH-ART 2012-001381-15; 2012-001381-15 (EudraCT Number)
Record Dates: First submitted 2012-08-02; First posted 2012-08-08 (Estimated); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Cystitis, Radio Induced
Keywords: Radio therapy; STRI; Urinary bladder; Hyperbaric Oxygen
MeSH Terms: conditions — Cystitis | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A - Immediate start (Active Comparator): Start of treatment within 6 weeks of inclusion in the study. 100% oxygen at 240-250 kPa will be delivered to the patents for 80-90 minutes while sitting or lying in a hyperbaric oxygen chamber. Patients will receive treatment once every day, except week-ends, for 40 days.
  Interventions: Drug: Hyperbaric Oxygen
- B - delayed start (No Intervention): Delayed start: Start of treatment not before 6 months of inclusion in the study. No intervention is given during the initial period.

INTERVENTIONS:
Drug: Hyperbaric Oxygen — 100% oxygen at 240-250 kPa will be delivered to the patents for 80-90 minutes while sitting or lying in a hyperbaric oxygen chamber. Patients will receive treatment once every day, except week-ends, for 40 days.
  Arms: A - Immediate start

SUMMARY:
The primary objective of this study is to assess the relief of symptoms after Hyperbaric Oxygen Therapy (HBOT) in patients with late radiation cystitis by having Expanded Prostate cancer Index Composite (EPIC)symptom estimation scale as primary variable.

Study hypothesis:

* HBOT can reduce or reverse the change or otherwise limit the damage of the bladder function and/or structure, which arose as a result of radiation therapy of cancer in the pelvic region organs.
* The effects of HBOT are associated with relief of symptoms that, at least in part, is related to the reduction of the extent of the radiation damage.
* Vascular density increases, fibrosis prevalence and inflammatory activity are reduced as a sign of an improved function of the mucosa.
* Treatment results of HBOT remains, in whole or in part, during the follow-up (residual effect)

DETAILED DESCRIPTION:
Radiotherapy is commonly used in the management of malignant diseases. Despite a continuous improvement of the technique, with improved efficacy and tolerance, adverse effects are still rather common. The urinary bladder and rectum are the major organs most commonly affected by radiotherapy to the pelvis area.

One of the most significant causes of the symptoms of radio therapy is inflammation and degeneration of blood vessels in the radiated tissue. Hyperbaric oxygen therapy involves administration of oxygen at greater than normal atmospheric pressures. A well-documented effect of HBOT is the stimulation of angiogenesis. HBOT is an established treatment for degeneration of blood vessels in the jaw bone as a result of radiotherapy and several publications have shown good efficacy also when soft tissue is affected.

If the method of treatment with HBOT means a reduction of the radiotherapy side effect it is thus an obvious importance for the individual patient. There is also significant potential savings for the healthcare and society.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures
* Female or male aged 18-80 years
* Intended curative radiation of the pelvic region as a treatment for cancer
* End of radiation therapy more than 6 months ago
* Radiation cystitis with Urological EPIC < 80
* Radiation cystitis is the most probable cause for the patient's symptoms

Exclusion Criteria:

* Patients with major and ongoing bleedings from the bladder (requiring more than 0.5L blood-transfusion within the last four weeks)
* Refractory incontinence requiring catheter or surgical intervention
* Urine bladder capacity < 100ml
* Fistula in the urine bladder
* Contraindications for HBOT according to the local centres routines
* Pregnancy
* Mechanical ventilator support
* Unable to follow and understand simple commands
* Not oriented to person, place and time

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2012-08; Primary Completion 2018-08-09 (Actual); Study Completion 2018-08-09 (Actual)

PRIMARY OUTCOMES:
EPIC (Expanded Prostate cancer Index Composite) | At inclusion, 6 months after inclusion (i.e. post treatment for group A and pre treatment for group B) and for long-term follow-up as specified under "description"
  EPIC was developed to measure health-related quality of life among men with prostate cancer (22) modified to enhance sensitivity to therapy effects. It comprises four summary domains; urinary, bowel, sexual and hormonal.
  The primary objective of this study is to assess the relief of symptoms after HBOT in patients with late radiation cystitis by having EPIC symptom estimation scale as primary variable, comparing results between group A (post treatment) and group B (pre treatment).
  All patients (Group A and B) will complete EPIC and SF-36 in a post-study long-term follow-up. This is done yearly for 5 years (18, 30, 42, 54 and 66 months post inclusion).

SECONDARY OUTCOMES:
Microscopic assessment | At inclusion and 6 months after inclusion (i.e. post treatment for group A and pre treatment for group B)
  To investigate the mucosa with respect to functionality by assessment of inflammation activity, quantification of fibrosis, vascular density and the presence of stems cells having histological analysis from biopsies as variable. Comparison will be made between group A (post treatment) and group B (pre treatment)
RTOG (Radiation Toxicity Grade by Radiation Therapy Oncology Group) | At inclusion and 6 months after inclusion (i.e. post treatment for group A and pre treatment for group B)
  RTOG is an internationally well established research group in the oncology field. They have developed organ specific scales for quantification of both acute and late symptoms after radiation. The scale range is from 0 to 5, where 0 is used for normal function and findings and 5 for death directly related to injuries post radiation. Both subjective and objective findings are used when setting the score.
  Comparison will be made between Group A (post treatment) and Group B (pre treatment)
SF-36 (Short Form Health Survey 36) | At inclusion, 6 months after inclusion (i.e. post treatment for group A and pre treatment for group B) and for long-term follow-up as specified under "description"
  SF-36 is a self-administered questionnaire and contains 36 items which measure eight dimensions and assess health-related quality of life. Comparing results between Group A (post treatment) and Group B (pre treatment).
  All patients (Group A and B) will complete EPIC and SF-36 in a post-study long-term follow-up. This is done yearly for 5 years (18, 30, 42, 54 and 66 months post inclusion).
Adverse events | Every day during HBOT (8 weeks).
  Adverse events (AE) are recorded during HBOT and Serious adverse events (SAE) until visit 4.

CONTACTS AND LOCATIONS:
Overall Officials: Nicklas Oscarsson, MD, Principal Investigator — Sahlgrenska, Gothenburg University
Locations (5):
- Rigshospitalet Copenhagen, Copenhagen, Denmark
- Turku Hospital, Turku, Finland
- Haukeland Universitetssykehus, Bergen, Norway
- Sweden (2):
  - Shalgrenska University Hospial, Gothenburg
  - Karolinska University Hospital, Stockholm

REFERENCES:
- [Derived] Oscarsson N, Rosen A, Muller B, Koskela LR, Giglio D, Kjellberg A, Ettala O, Seeman-Lodding H. Radiation-induced cystitis treated with hyperbaric oxygen therapy (RICH-ART): long-term follow-up of a randomised controlled, phase 2-3 trial. EClinicalMedicine. 2025 Apr 19;83:103214. doi: 10.1016/j.eclinm.2025.103214. eCollection 2025 May. PMID 40291346
- [Derived] Oscarsson N, Muller B, Rosen A, Lodding P, Molne J, Giglio D, Hjelle KM, Vaagbo G, Hyldegaard O, Vangedal M, Salling L, Kjellberg A, Lind F, Ettala O, Arola O, Seeman-Lodding H. Radiation-induced cystitis treated with hyperbaric oxygen therapy (RICH-ART): a randomised, controlled, phase 2-3 trial. Lancet Oncol. 2019 Nov;20(11):1602-1614. doi: 10.1016/S1470-2045(19)30494-2. Epub 2019 Sep 16. PMID 31537473

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-05-15): https://cdn.clinicaltrials.gov/large-docs/23/NCT01659723/SAP_000.pdf
  • Study Protocol and Informed Consent Form (2014-05-01): https://cdn.clinicaltrials.gov/large-docs/23/NCT01659723/Prot_ICF_001.pdf